CLINICAL TRIAL: NCT02689349
Title: Esteem Totally Implantable Hearing System New Subject Enrollment Post Approval Study
Brief Title: Esteem New Subject Enrollment Post Approval Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Envoy Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0205
Record Dates: First submitted 2016-02-08; First posted 2016-02-23 (Estimated); Results first posted 2022-06-01 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Sensorineural Hearing Loss
Keywords: hearing; implant; moderate degree; severe degree
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Esteem Implant Prospective Subjects (Experimental): Subjects followed through 1 year for both Safety and Efficacy endpoints
  Interventions: Device: Implantation of Esteem
- Esteem Implant Retrospective Chart Review Subjects (Other): Subjects providing Safety-only endpoint data through retrospective chart review, to be added to Prospective Subjects' Safety data
  Interventions: Device: Implantation of Esteem

INTERVENTIONS:
Device: Implantation of Esteem — Subjects meeting indications are implanted with the Esteem Totally Implantable Hearing System

SUMMARY:
The New Enrollment Post-Approval Study is designed to evaluate the safety and efficacy of the Esteem Totally Implantable Hearing System in subjects suffering from moderate to severe hearing loss.

DETAILED DESCRIPTION:
Purpose:

To evaluate the long-term safety and efficacy of the Esteem Totally Implantable Hearing System (hereafter called Esteem) in subjects suffering from moderate to severe hearing loss.

Questions:

The following questions are to be answered:

* Is Esteem effective through 1 year follow-up?
* Is Esteem safe through 1 year follow-up?
* Is the incidence of facial paresis/paralysis at 1 month follow-up no greater than 7%?

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years old
2. Subject understands the nature of the procedure and has signed the Subject Informed Consent Form prior to the procedure
3. Subject is willing and able to comply with specified follow-up evaluations and understands the audiological test procedures and use of the Esteem® System.
4. Subject has moderate to severe sensorineural hearing loss in the ear to be implanted defined by pure tone average air-conduction threshold level.
5. Subject has an unaided maximum word recognition score of greater than or equal to 40% with recorded delivery using a phonetically balanced word list at SRT + 40 decibels (dB) or at maximum tolerable presentation level.
6. Subject is a current user of a properly functioning and appropriately fit hearing aid for at least one (1) month in the ear to be implanted.
7. Subject has normally functioning eustachian tube
8. Subject has normal tympanic membrane
9. Subject has a normal middle ear anatomy
10. Subject has adequate space for Esteem® System implant determined via fine cut temporal bone CT scan
11. Subject is a native speaker of the English language.

Exclusion Criteria:

1. Subject has a history of post-adolescent chronic middle ear infections, inner ear disorders or recurring vertigo requiring treatment, disorders such as mastoiditis, Hydrops or Meniere's syndrome or disease
2. Subject has a history of otitis externa or eczema for the outer ear canal and the investigator believes this will affect the Esteem® System implantation
3. Subject has cholesteatoma or destructive middle ear disease
4. Subject has life expectancy of < two (2) years due to other medical conditions
5. Subject has retrocochlear or central auditory disorders
6. Subject is known to be suffering from any psychological, developmental, physical, or emotional disorder that the investigator feels would interfere with the surgery or follow-up testing
7. Subject has a known history of fluctuating air conduction and/or bone conduction hearing loss over a one-year period of 15 dB in either direction at 2 or more frequencies (from 500 - 4000 Hz)
8. Subject has sudden hearing loss due to unknown cause
9. Subject has a history of disabling tinnitus, defined as tinnitus which required treatment.
10. Subject is unable to adequately perform audiological testing
11. Subject has a medical condition or undergoing a treatment that may affect healing and the investigator does not believe the subject is a good candidate for the trial.
12. Subject has diabetes that is not well controlled with medication or diet and the investigator does not believe in his best medical judgment that the subject would be a good candidate for the trial
13. Subject is pregnant at the time of device implant
14. Subject has a history of keloid formation
15. Subject has known hypersensitivity to silicone rubber, polyurethane, stainless steel, titanium and/or gold

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sam Marzo, MD, Principal Investigator — Loyola Center for Hearing, Woodridge IL; John Li, MD, Principal Investigator — Jupiter Medical Center, Jupiter FL; Deborah Clark, AuD, Principal Investigator — Pacific Hearing Service, Los Altos CA; Wayne Berryhill, MD, Principal Investigator — Oklahoma Otolaryngology Associates; Sanjay Bhansali, MD, Principal Investigator — Ear Consultants of Georgia; Abraham Jacob, MD, Principal Investigator — University of Arizona Ear Institute; Elizabeth Toh, MD, Principal Investigator — Lahey Hospital & Medical Center
Locations (6):
- United States (6):
  - North Alabama ENT Associates, Madison, Alabama
  - Pacific Hearing Service, Los Altos, California
  - Ear, Nose, & Throat Associates of South Florida, Jupiter, Florida
  - Ear Consultants of Georgia, Atlanta, Georgia
  - Loyola Center for Hearing, Woodridge, Illinois
  - Oklahoma Otolaryngology Associates, Norman, Oklahoma

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Esteem Implant Prospective Subjects: Implantation of Esteem: Subjects meeting indications are implanted with the Esteem Totally Implantable Hearing System and followed for both Efficacy and Safety endpoints.
- Esteem Implant Retrospective Chart Review Subjects: Subjects whose clinical data (Safety only) were obtained retrospectively to achieve required N for Safety endpoints
Period: Overall Study
Arm/Group | Esteem Implant Prospective Subjects | Esteem Implant Retrospective Chart Review Subjects
Started | 59 | 58
Completed | 46 | 58
Not Completed | 13 | 0
Not completed — Not implanted | 4 | 0
Not completed — Withdrawal by Subject | 9 | 0

BASELINE CHARACTERISTICS:
Groups:
- Esteem Implant Prospective Subjects: Subjects meeting indications for candidacy are followed through 1 year for both Safety and Efficacy endpoints
- Esteem Implant Retrospective Chart Review Subjects: Subjects meeting indications for candidacy for Safety endpoints provide Safety-only data via retrospective chart review, which will supplement the Prospective Subjects' Safety data in order to reach required N.
- Total: Total of all reporting groups
Arm/Group | Esteem Implant Prospective Subjects | Esteem Implant Retrospective Chart Review Subjects | Total
Number analyzed (Participants) | 59 | 58 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Demographic data were not collected on Retrospective Chart Review subjects.
  years
    number analyzed (Participants) | 59 | 0 | 59
    (all) | 60.4 (17.6) |  | 60.4 (17.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Demographic data were not collected on Retrospective Chart Review subjects Population: Demographic data were not collected on Retrospective Chart Review subjects.
  Participants
    number analyzed (Participants) | 59 | 0 | 59
    Female | 17 | 0 | 17
    Male | 42 | 0 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Baseline data were not collected on Retrospective Chart Review subjects
  Participants
    White/Caucasian: number analyzed (Participants) | 59 | 0 | 59
    White/Caucasian | 58 |  | 58
    Black/Non-Hispanic: number analyzed (Participants) | 59 | 0 | 59
    Black/Non-Hispanic | 1 |  | 1
    Hispanic: number analyzed (Participants) | 59 | 0 | 59
    Hispanic | 0 |  | 0
    Asian: number analyzed (Participants) | 59 | 0 | 59
    Asian | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 59 | 58 | 117
Work status [Count of Participants; unit: Participants] — Describes reported work status of participant, whether working full-time, part-time, retired, or unemployed. Population: Demographic data were not collected on subjects in retrospective chart review cohort.
  Participants
    work full-time: number analyzed (Participants) | 59 | 0 | 59
    work full-time | 17 | 0 | 17
    work part-time: number analyzed (Participants) | 59 | 0 | 59
    work part-time | 6 | 0 | 6
    retired: number analyzed (Participants) | 59 | 0 | 59
    retired | 24 | 0 | 24
    unemployed: number analyzed (Participants) | 59 | 0 | 59
    unemployed | 3 | 0 | 3
    other: number analyzed (Participants) | 59 | 0 | 59
    other | 7 | 0 | 7
    did not answer: number analyzed (Participants) | 59 | 0 | 59
    did not answer | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Speech Reception Threshold (SRT)
Description: Comparison of the speech reception threshold (SRT) using the Esteem System as compared to the pre-implant aided condition. The SRT is related to hearing sensitivity; lower numbers indicate better outcomes. Here, the difference in dB is reported; positive scores indicate improvement (lower SRT) with the Esteem relative to the pre-implant hearing aid. There are no specific minimum or maximum scores for this measure.
Time Frame: Change in SRT from Baseline Aided to 10-month post-activation with Esteem
Population: Change in Speech Reception Threshold (SRT) was not collected from the Esteem Implant Retrospective Chart Review Subject Arm.
Measure: Mean (Standard Error); unit: dB
Groups:
- Esteem Implant Prospective Subjects: Subjects meeting indications are implanted with the Esteem Totally Implantable Hearing System and followed for both Safety and Efficacy endpoints for 1 year.
Arm/Group | Esteem Implant Prospective Subjects
Number analyzed (Participants) | 46
dB | 5.3 (2.4)

2. Primary Outcome: Change in Word Recognition Score (WRS)
Description: Comparison of the word recognition score using the Esteem compared to the pre-implant aided condition. For WRS, a higher score indicates a better outcome. Here, the difference in % correct is reported; positive scores indicate better performance with the Esteem relative to the pre-implant hearing aid. Scores on this test range from 0 to 100%.
Time Frame: Change in WRS from Baseline Aided to 10-month post-activation with Esteem
Population: Change in Word Recognition Score (WRS) was not collected from the Esteem Implant Retrospective Chart Review Subject Arm.
Measure: Mean (Standard Error); unit: percent correct
Arm/Group | Esteem Implant Prospective Subjects
Number analyzed (Participants) | 46
percent correct | 5.5 (3.8)

3. Primary Outcome: Incidence of SADEs, Device Failures, & Replacements
Description: The analysis of the incidence of Serious Adverse Device Effects (SADEs) and device failures and replacements
Time Frame: Incidence at 10-month post-activation
Measure: Number; unit: Number of events
Arm/Group | Esteem Implant Prospective Subjects | Esteem Implant Retrospective Chart Review Subjects
Number analyzed (Participants) | 46 | 58
Number of events | 3 | 0

4. Primary Outcome: Incidence of Facial Pareses/Paralysis
Description: The analysis of the incidence of facial pareses/paralysis at one month follow-up
Time Frame: Incidence at one month post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Esteem Implant Prospective Subjects | Esteem Implant Retrospective Chart Review Subjects
Number analyzed (Participants) | 46 | 58
Participants | 3 | 0

5. Primary Outcome: Change in Bone Conduction Threshold (BCT) at 500 Hz
Description: Comparison of bone conduction (BC) threshold at 500 Hz post activation compared to the pre-implant BC threshold. Change in Bone Conduction is used to determine whether residual cochlear function has declined following implant of the Esteem. Positive numbers indicate higher (i.e., poorer) bone conduction thresholds post-implant, relative to pre-implant.
Time Frame: Change in BCT from Baseline to 10-month post-activation
Population: Change in Bone Conduction Threshold (BCT) at 500 Hz was not collected from the Esteem Implant Retrospective Chart Review Subject Arm.
Measure: Mean (Standard Error); unit: dB
Arm/Group | Esteem Implant Prospective Subjects
Number analyzed (Participants) | 46
dB | 1.4 (2.0)

6. Primary Outcome: Change in Bone Conduction Threshold (BCT) at 1000 Hz
Description: Change in BCT from Baseline to 10-month post-activation. Change in Bone Conduction is used to determine whether residual cochlear function has declined following implant of the Esteem. Positive numbers indicate higher (i.e., poorer) bone conduction thresholds post-implant, relative to pre-implant.
Time Frame: Change in BCT from Baseline to 10-month post-activation
Population: Change in Bone Conduction Threshold (BCT) at 1000 Hz was not collected from the Esteem Implant Retrospective Chart Review Subject Arm.
Measure: Mean (Standard Error); unit: dB
Arm/Group | Esteem Implant Prospective Subjects
Number analyzed (Participants) | 46
dB | 1.8 (2.2)

7. Primary Outcome: Change in Bone Conduction Threshold (BCT) at 2000 Hz
Description: as for outcome 6
Time Frame: Change in BCT from Baseline to 10-month post-activation
Population: Change in Bone Conduction Threshold (BCT) at 2000 Hz was not collected from the Esteem Implant Retrospective Chart Review Subject Arm.
Measure: Mean (Standard Error); unit: dB
Arm/Group | Esteem Implant Prospective Subjects
Number analyzed (Participants) | 46
dB | 2.3 (2.7)

8. Primary Outcome: Change in Bone Conduction Threshold (BCT) at 4000 Hz
Description: as for outcome 6
Time Frame: Change in BCT from Baseline to 10-month post-activation
Population: Change in Bone Conduction Threshold (BCT) at 4000 Hz was not collected from the Esteem Implant Retrospective Chart Review Subject Arm.
Measure: Mean (Standard Error); unit: dB
Arm/Group | Esteem Implant Prospective Subjects
Number analyzed (Participants) | 46
dB | -3.4 (2.0)

9. Secondary Outcome: Change in Subjective Quality of Life as Measured With the Abbreviated Profile of Hearing Aid Benefit, or APHAB (Global Score)
Description: Quality of Life measured with the APHAB comparison between the pre-implant aided condition and 10-month post-activation. In general, a lower score indicates better performance. The range of scores for each subscale (including the Global score, reported here) is 1 to 99. Here, mean difference in benefit score with the Esteem implant vs. pre-implant aided condition is reported. A positive difference score indicates more benefit with the Esteem.
Time Frame: Change from Baseline Aided to 10-month post-activation with Esteem
Population: Questionnaire data available from only 41 of 46 subjects. The APHAB (Global Score) was not collected from the Esteem Implant Retrospective Chart Review Subject Arm.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Esteem Implant Prospective Subjects
Number analyzed (Participants) | 41
score on a scale | 5.8 (3.1)

10. Secondary Outcome: Esteem Questionnaire Results
Description: To gather subject feedback and comments on the use of the Esteem System through subject ratings on questionnaire items specifically focusing on factors such as the clarity of sound, the user's ability to understand speech in background noise, naturalness of sound, benefits of the system, etc. -- relative to the pre-implant aided condition. Subjects rated each item as "Is much worse", "Somewhat worse", "Is about the same", "Is somewhat better", or "Is much better" with the Esteem. Reported here are the cumulative number of respondents indicating "Same", "Somewhat better", or "Much better" for the given question.
Time Frame: 10-month post-activation with Esteem
Population: Esteem Questionnaire Results were not collected from the Esteem Implant Retrospective Chart Review Subject Arm. Three subjects did not complete the Esteem Questionnaire at the 10-month visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Esteem Implant Prospective Subjects
Number analyzed (Participants) | 43
Participants
  1. How do you rate the clarity of the sound you hear with the Esteem compared to your hearing aid? | 37
  How do you rate your ability to understand speech in background noise ... ? | 33
  How natural sounding are voices and other sounds compared to your hearing aid? | 36
  How do you rate the benefit of the entire system being invisible ... compared to your hearing aid? | 36
  How well do you understand conversation with your Esteem even when several people are talking ...? | 38
  How confident do you feel with the Esteem compared to your hearing aid? | 41
  Does the Esteem allow you to live a more active lifestyle? | 43

ADVERSE EVENTS:
Time Frame: Adverse events reported here were those occurring within 10 months post-implantation
Description: Adverse Event (AE): any undesirable clinical event occurring to a subject, during a clinical trial, whether or not it is considered related to the investigational product.
  Serious Adverse Event (SAE) or Serious Adverse Device Effect (SADE): any adverse event that results in death, is life threatening, is disabling, involves cancer or congenital anomaly, requires or prolongs in-patient hospitalization (>24 hours) and/or requires intervention to prevent permanent impairment / damage.
Groups:
- Esteem Implant Prospective Subjects: Subjects meeting indications who were implanted with the Esteem Totally Implantable Hearing System and followed for both Efficacy and Safety endpoints.
Arm/Group | Esteem Implant Prospective Subjects | Esteem Implant Retrospective Chart Review Subjects
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/58
Serious Adverse Events (participants affected / at risk) | 9/59 | 0/58
Other Adverse Events (participants affected / at risk) | 23/59 | 5/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esteem Implant Prospective Subjects (N=59) | Esteem Implant Retrospective Chart Review Subjects (N=58)
Fibrotic tissue in middle ear (Ear and labyrinth disorders) | 3 (3) | 0 (0) — Adjudicated as moderate procedure-related SAE in three cases, moderate device-related AE in one case, and as severe SADE in one case.
Facial weakness/paresis (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) — Procedure-related SAE, mild in one case and moderate in two cases.
Incision breakdown (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Adjudicated as procedure-related SAE of moderate severity.
Silicone erosion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Adjudicated as moderate device-related SAE
Infection (Infections and infestations) | 1 (1) | 0 (0) — Adjudicated as moderate procedure-related SAE
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esteem Implant Prospective Subjects (N=59) | Esteem Implant Retrospective Chart Review Subjects (N=58)
Incision discomfort (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — Adjudicated as mild procedure-related AE
Taste disturbance (Injury, poisoning and procedural complications) | 17 (17) | 1 (1) — Adjudicated as mild procedure-related AE
Uncomfortable sound (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Adjudicated as mild device-related AE.
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Adjudicated as mild AE
Numbness (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) — Adjudicated as mild procedure-related AE
Air bubble over implant (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) — Adjudicated as mild procedure-related AE
Device cuts out (Ear and labyrinth disorders) | 1 (1) | 1 (1) — Adjudicated as procedure-related AE
Disequilibrium (Ear and labyrinth disorders) | 2 (2) | 0 (0) — Adjudicated as mild, procedure-related AE
Tinnitus (Ear and labyrinth disorders) | 6 (6) | 0 (0) — Adjudicated as mild AE
Noise or audible artifact (Ear and labyrinth disorders) | 2 (2) | 0 (0) — Adjudicated as mild AE
Clarity or sound quality (Ear and labyrinth disorders) | 2 (2) | 0 (0) — Adjudicated as mild, device-related AE
Suction feeling at implant site (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Adjudicated as moderate, procedure-related AE
Non-implant hearing aid sound quality (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Adjudicated as mild AE
Lump at implant site (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Adjudicated as mild device-related AE
Fell and hit head (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Adjudicated as moderate AE
Middle ear effusion (Ear and labyrinth disorders) | 3 (3) | 0 (0) — Adjudicated as mild, procedure-related AE in two cases, and moderate, procedure-related AE in one case.
Ear drainage (Ear and labyrinth disorders) | 2 (2) | 0 (0) — Adjudicated as mild, procedure-related AE.
Keloids (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Adjudicated as mild, procedure-related AE
Incision breakdown (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Adjudicated as mild, procedure-related AE
High capacitance measurement (Product Issues) | 0 (0) | 1 (1) — Device-related AE
Personal Programmer malfunction (Product Issues) | 0 (0) | 1 (1) — Device-related AE
Limited benefit (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Based on post-market surveillance complaint. Per site, "resolved with medication - no device deficiency noted."

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT02689349/Prot_SAP_000.pdf